CLINICAL TRIAL: NCT03663881
Title: Open-label, Single Arm, Phase 1 Study to Assess the Safety of P2Et Extract Obtained From Caesalpinia Spinosa, in Voluntary Subjects in Colombia
Brief Title: Safety Assessment of P2Et Extract in Healthy Voluntary Subjects in Colombia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS001-SA
Record Dates: First submitted 2018-08-08; First posted 2018-09-10 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Toxicity; Safety Issues
Keywords: Polyphenols; Safety; Herbal Extract

STUDY DESIGN:
Intervention Model Description: Open-label, single arm, Phase 1 study. 24 participants are anticipated, assuming that 6 participants are recruited in each of the levels of dose titration based on the 3 +3 design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- P2Et extract (Experimental): P2Et extract daily doses. Dosage scaling will be performed according to the 3 + 3 standard design.
  Interventions: Drug: P2Et extract

INTERVENTIONS:
Drug: P2Et extract — P2Et extract daily doses. Dosage scaling will be performed according to the 3 + 3 standard design.
  Other Names: P2Et obtained from Caesalpinia spinosa

SUMMARY:
Caesalpinia spinosa extract is rich in gallotannins and other well characterized polyphenols and has a major antioxidant activity. The extract shows immunomodulatory activity in healthy animals and anti-tumor activity in animals with breast cancer and melanoma as well.

The use of P2Et in animals with tumors shows a synergistic effect with doxorubicin in drug-resistant cell lines. In addition, an increase in survival of transplanted animals with a TS/A breast cancer tumor model and treated with P2Et, in conjunction with calreticulin increase is observed.

This open-label, single arm, Phase 1 study intends to assess the safety of P2Et extract obtained from Caesalpinia spinosa, with dose escalation, in healthy voluntary participants in Colombia.

DETAILED DESCRIPTION:
The P2Et extract will be self-administered by the participants on a daily basis (600 mg 1 daily capsule, 2 daily capsules for 1,200 mg, 4 daily capsules for 2,400 and 8 daily capsules for 4,800 mg) 1 hour after meals and at the same time every day, from day 1 to day 30.

In the event that the participants presents vomit within 15 minutes after taking P2Et, the participants should take another dose. Should the participant forget any scheduled dose and less than 6 hours have elapsed, the participant must take the dose immediately; if more than 6 hours have elapsed, the subject must wait and take the next scheduled dose.

Dose escalation will be performed to determine the P2Et maximum tolerated dose (MTD) and maximum dose toxicity (MDT). In the escalation phase, the P2Et daily dose will be escalated in the cohort of subjects with minimum dose of 600 mg daily to a maximum of 4,800 mg. Each cohort will be made up of around 3 and 6 subjects, at least 3 subjects will be enrolled in each dosage level. Should MTD is not observed in the first 3 subjects treated in the first month, escalation to the next dosage level will be undertaken. Should 1 or more MTD occur in any dosage level in a subject, 3 subjects will be added to that cohort.

Any dosage level in which 2 out of 6 subjects experience a MTD will be considered intolerable and the previous dose will be considered the P2Et maximum tolerated dose (MTD) and dose escalation will be terminated. The 3+3 design will be used monthly for the P2Et dose escalation (up to a maximum of 4.8 g/day).

The participants will be followed-up until withdrawal of the protocol therapy. The participants removed from the protocol due to unacceptable adverse events will be followed-up until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Adequate renal, hematological, hepatic function defined as:

   * Normal renal function defined as serum creatinine ≤ 1.5 mg/dl or creatinine clearance

     * 60 mL/min/1.73 m2 (according to local evaluation method).
   * Hepatic function: alkaline phosphatase ≤ 2.5 × LSN, aspartate aminotransferase (AST) ≤ 2.5 × LSN, alanine aminotransferase ≤ 2.5 × LSN, total bilirubin ≤ 1.5 × LSN.
   * Leukocyte count ≥3,000/mcL, neutrophils absolute count ≥ 1500/mm3 (1.5 × 109/L).

   Platelets ≥100,000/mm3 (100 × 109/L) and Hemoglobin ≥ 9.0 g/dL in peripheral blood.

   - Cardiovascular function: No evidence of acute ischemic heart disease in the electrocardiogram.
3. No uncontrolled or significant comorbidities determined by clinical history, physical examination and screening laboratory tests at the discretion of the investigator.
4. Women of childbearing age must have a negative pregnancy test (urine or serum) at the time of screening and enrollment.
5. Female subjects of childbearing age (those who have not been menopausal at least for 12 months or who have undergone surgical sterilization by bilateral tubal ligation procedure, bilateral oophorectomy or hysterectomy), and their male partners, must use at least one of the below mentioned contraceptive methods at the time of entering the study, throughout the study, and at least 6 months following the P3Et use (the effects of

   P2Et in the developing human fetus are unknown):
   1. Total abstinence of sexual intercourse, starting at least one complete menstrual cycle prior to the administration of the study drug; (it should be noted that: sexual abstinence as a contraceptive method must be limited to those cases in which it has been established as the pre-existent election of lifestyle by the patient);
   2. Vasectomized partner of a female subject.
   3. Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to the administration of the study drug;
   4. Intrauterine device (IUD)
   5. Double barrier method (condom, contraceptive sponge, diaphragm or vaginal ring with spermicidal gel or foam).
6. Willingness to complete the study interventions and follow-up.
7. The subject must sign and date the informed consent form voluntarily for his (her) participation in the study, approved by an Institutional Ethics Committee (IEC) prior to the initiation of any selection procedure or specific to the study.

Exclusion Criteria:

Subjects with one or more of the following conditions are not eligible for this study.

1. Subjects receiving any investigational agent and /or taking part in a clinical study in the 30 days prior to the admission or during their participation in the study.
2. History of allergic reactions attributed to polyphenol-type compounds similar to those found in green tea.
3. Use of dietary supplements or phytopharmaceutical drugs < 15 days prior to the admission and during the study.
4. Subjects with diagnosis of an active disease and/or receiving pharmacological treatment prescribed for an active disease and who have evidence of an active disease at the time of the initial clinical examination at the discretion of the investigator.
5. Severe, active concomitant morbidity, including but not limited to:

   * Bacterial or fungal acute infection requiring intravenous antibiotics at the time of inclusion.
   * Moderate or severe liver failure (B or higher Child-Pugh category with qualification 7 or higher).
   * Congestive heart failure grade II or higher according to New York Heart Association requiring hospitalization within 12 months prior to registration.
   * Unstable angina and/or congestive heart disease within the previous 6 months
   * Severe cardiac arrhythmia with no appropriate control.
   * Antecedents of brain hemorrhage or stroke (ACV) or transient ischemic attack within the previous 6 months.
   * Myocardial infarction within the previous 6 months.
   * Exacerbation of chronic obstructive pulmonary disease or another respiratory disease requiring hospitalization or that precludes the study treatment at the time of inclusion.
   * Subjects with a disease indicative of clinically defined Acquired Immunodeficiency Syndrome (AIDS). This is necessary in order to assure that those subjects can be more likely to be suitable to receive the full treatment.
   * Any other major clinical disease or psychiatric disorder that, at the discretion of the investigator, precludes the administration or completion of the protocol treatment.
6. Voluntary subjects having history or drugs and/or alcohol abuse.
7. Voluntary subjects who are smokers at the time of the screening visit.
8. Subjects who have received strong or moderate CYP3A inductors and inhibitors listed in the Appendix A within 7 days prior to the treatment initiation.
9. The female subject is pregnant or breastfeeding.

   * Bacterial or fungal acute infection requiring intravenous antibiotics at the time of inclusion.
   * Moderate or severe liver failure (B or higher Child-Pugh category with qualification 7 or higher).
   * Congestive heart failure grade II or higher according to New York Heart Association requiring hospitalization within 12 months prior to registration.
   * Unstable angina and/or congestive heart disease within the previous 6 months.
   * Severe cardiac arrhythmia with no appropriate control.
   * Antecedents of brain hemorrhage or stroke (ACV) or transient ischemic attack within the previous 6 months.
   * Myocardial infarction within the previous 6 months.
   * Exacerbation of chronic obstructive pulmonary disease or another respiratory disease requiring hospitalization or that precludes the study treatment at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 12 months
  Identification of the maximum dose toxicity

SECONDARY OUTCOMES:
Immunomodulation | 12 months
  Change between baseline immunological profile percentage and end of the treatment immunological profile percentage with its respective mean, median, standard deviation and range.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Torregrosa Almonacid, MD, Principal Investigator — Surgeon
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Colombia